CLINICAL TRIAL: NCT00760630
Title: Simultaneous Measurements of Pressure Gradient, Blood Flow and Percentage Area Stenosis of Coronary Epicardial Lesions to Assess Severity of Epicardial Stenosis and Myocardial Infarction
Brief Title: Measurements to Assess Severity of Epicardial Stenoses
Acronym: MASES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB Approval expired on 05/28/09 as it was pilot study. A new study was later initiated once VA Merit Review Grant (I01CX000342-01) was received. Thus a new IRB (10-05-05-02) and clinicaltrials.gov (NCT01719016) were initiated in place of this study.
Sponsor: University of Cincinnati (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Rupak K. Banerjee, Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UCIRB08031108
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
Keywords: abnormal stress test; fractional flow reserve; pressure drop coefficient; lesion flow coefficient
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CDP LFC (Experimental): all patients will have this calculation based upon diagnostic parameters with IVUS and FFR and/or CFR
  Interventions: Device: FFR/CFR and IVUS

INTERVENTIONS:
Device: FFR/CFR and IVUS — All patients with clinical indication for cardiac cath will have FFR and IVUS
  Other Names: Volcano FFR and IVUS catheters will be used

SUMMARY:
Newly developed diagnostic parameters have potential to differentiate between epicardial disease and microvascular dysfunction with the help of anatomical details and physiological endpoints and can be used in present clinical settings.

DETAILED DESCRIPTION:
The pressure drop coefficient (CDP) is a functional index based on hyperemic dp and u measurements. The lesion flow coefficient (LFC) combines the functional index CDP with an atomic measure (percentage area stenosis) as a single parameter.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal Myocardial stress perfusion (SPECT) LV EF > 25%

Exclusion Criteria:

* LV < or + to 25% Serum Creatinine > 2.5 gm/dL Type II HIT Significant co-morbidities Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2012-02-24 (Actual); Study Completion 2012-02-24 (Actual)

PRIMARY OUTCOMES:
to detect ischemic heart disease in patients with abnormal stress tests using MPI with SPECT and to determine the presence of significant epicardial stenosis using coronary angiography with simultaneous physiological pressure and flow measurements | Upon Diagnostic Angiogram and Flow Wire

SECONDARY OUTCOMES:
To compare novel measurements, Pressure Drop Coefficient (CDP) & Lesion Flow Coefficient (LFC), against measured current parameters called Fractional flow reserve (FFR) & Coronary flow reserve (CFR). | Upon Diagnostic Angiogram and Flow Wire

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Effat, MD, Principal Investigator — University of Cincinnati; Kranthi K Kolli, MS, Principal Investigator — University of Cincinnati; Massoud Leesar, MD, Principal Investigator — University of Cincinnati; Rupak Banerjee, PhD, Principal Investigator — University of Cincinnati; Tarek Helmy, MD, Principal Investigator — University of Cincinnati; Srikara Pellukhana, BS, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - University Hospital, Cincinnati, Ohio
  - Department of Veterans Affairs, Cincinnati, Ohio